CLINICAL TRIAL: NCT02905721
Title: Evaluation of Spectral Cardiac CT for the Diagnosis of Acute Myocarditis
Acronym: MYOCARDITESCAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AOM 150399 / P 150927
Record Dates: First submitted 2016-09-07; First posted 2016-09-19 (Estimated); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Patients With Suspected Acute Myocarditis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spectral cardiac CT scan (Experimental): All patients will undergo cardiac CT scan with spectral mode acquisition
  Interventions: Procedure: Spectral cardiac CT scan

INTERVENTIONS:
Procedure: Spectral cardiac CT scan — Cardiac CT scan : acquisition using the spectral mode imaging in order to identify inflammatory areas of the myocardium on the iodine map imaging.

SUMMARY:
Spectral cardiac CT scan performed in an emergency setting in patients with suspected acute myocarditis and presenting one selves with an acute chest pain, allows the non-invasive assessment of both the coronary arteries and the myocardium. Delayed iodine contrast-enhanced CT imaging should show the inflamed area with an increased uptake of iodine contrast agent in the interstitial space, such as the well-known hypersignal seen on the myocardial delayed enhancement sequence with MRI (corresponding of an uptake of gadolinium contrast agent in the abnormal myocardium).

This technique has the potential to replace MRI, thus allowing the diagnosis of acute myocarditis with a rapid and easily accessible technique. Moreover, it has the additional benefit of avoiding invasive coronary angiography in the specific population of patients without any significant risk factors of atheromatous disease.

DETAILED DESCRIPTION:
Introduction: diagnosis of acute myocarditis is challenging in the specific population of patients without any significant risk factors of atheromatous disease.

Both cardiac MRI and coronary angiography (cardiac CT, invasive coronary angiography) are usually performed for the definitive diagnosis of myocarditis and for ruling out a coronary artery disease.

Spectral cardiac CT could be particularly useful in suspected myocarditis in the setting of acute chest pain in this specific population of patients with low cardiovascular risk factors. Indeed, both coronary arteries and myocardial tissue can be assessed on the same technique (cardiac CT scan) which offers the advantages of being non-invasive, more available and more easily used than MRI in emergency situations. Cardiac CT allows the detection of abnormal myocardial territories by showing subepicardial iodinated contrast enhancement with the spectral mode imaging. It also allows the direct visualization of coronary arteries, thus preventing the necessity of performing coronary angiography in a significant number of patients with suspected myocarditis in the setting of acute chest pain.

Primary objective: to evaluate the diagnostic accuracy of spectral cardiac CT imaging for the diagnosis of acute myocarditis using cardiac MRI as the gold standard, in patients with suspected myocarditis in the setting of acute chest pain. The diagnosis of acute myocarditis using spectral cardiac CT scan will be based on the presence of late subepicardial contrast enhancement detected using iodine imaging obtained after subtraction of water imaging. The gold standard will be the diagnosis of acute myocarditis based on the state-of-the-art MRI criteria.

Secondary objective: to assess the radiation dose delivered in spectral cardiac CT scan using the latest generation of machines from different manufacturers (such as GE Healthcare and Siemens).

Experimental plan: Multicenter diagnostic accuracy study, conducted within the scope of routine care of patients admitted for suspected acute myocarditis, conducted according to the Standards for the Reporting of Diagnostic (STARD) guidelines. Clinical, laboratory, cardiac MRI, and invasive coronary angiography are performed in routine care. Cardiac MRI serves as the reference standard for the definitive diagnosis of acute myocarditis. Cardiac CT is also performed in routine care in order to rule out a coronary disease. The investigators will add a second acquisition using the spectral mode imaging in order to identify inflammatory areas of the myocardium on the iodine map imaging.

All patients will undergo both cardiac CT scan with spectral mode acquisition and cardiac MRI to avoid work-up bias. Spectral CT imaging and cardiac MRI will be performed within 72 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged at least 18 years
* Patient having had a preliminary clinical examination:

eligible patients must present an increased level of troponin I (>laboratory threshold) associated with at least one of the 3 following criteria: i) prolonged chest pain > 10 minutes; ii) recent viral infectious illness <7 days; iii) patients without any history of coronary disease and/or free of cardiovascular risk factors

- Patient's written informed consent.

Exclusion Criteria:

* Iodine contrast allergy
* Severe renal impairment (GFR < 45 ml/min)
* Patient status: insufficient patient cooperation or dyspnea or hemodynamic instability with inability to hold a 8-10 seconds breath hold
* Pregnant women
* History of coronary artery disease
* Contra indications to MRI
* Patient under guardianship or trusteeship
* Non affiliation to social security or CMU (beneficiary or assignee)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2017-10-11 (Actual); Primary Completion 2022-10-10 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of acute myocarditis using spectral cardiac CT scan | 72 hours
  The test under study is the spectral cardiac CT scan. Diagnosis of acute myocarditis using spectral cardiac CT scan will be based on the presence of a contrast enhancement involving the subepicardial layers of the myocardial.

SECONDARY OUTCOMES:
Radiation dose delivered in spectral cardiac CT scan | 72 hours
  The radiation dose delivered in spectral cardiac CT scan using the latest generation of machines from different manufacturers (GE Healthcare and Siemens)

CONTACTS AND LOCATIONS:
Overall Officials: Phalla OU, MD PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Bichat Claude Bernard Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided